CLINICAL TRIAL: NCT07254858
Title: Combined Chemo-immunotherapy Plus SBRT in Neoadjuvant Treatment for Luminal Subtype Breast Cancer: A Prospective Multicenter Randomized Controlled Trial
Brief Title: Combined Chemo-immunotherapy Plus SBRT in Neoadjuvant Treatment for Luminal Subtype Breast Cancer
Acronym: CISN-L
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Wang Ouchen, Chief Physician, First Affiliated Hospital of Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2025-301
Record Dates: First submitted 2025-09-08; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-09

CONDITIONS: HR+/HER2- Breast Cancer
Keywords: Breast Cancer; Radiotherapy; Immunotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Neoadjuvant Therapy; Immunotherapy; sintilimab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chemotherapy+Immunotherapy (Experimental): Control Group: Neoadjuvant chemotherapy combined with immunotherapy, wherein the neoadjuvant chemotherapy regimen follows the clinical standard protocol.
  Neoadjuvant Chemotherapy Regimen:
  A sequential chemotherapy strategy is adopted, with the specific regimen as follows:
  Taxane-based Chemotherapy Phase (T Phase):
  Nab-paclitaxel (125 mg/m²), administered by intravenous infusion on Day 1 and Day 8 of each 21-day cycle (Q3W), for a total of 4 cycles.
  Anthracycline-based Combination Chemotherapy Phase (EC Phase):
  Epirubicin (75-100 mg/m²) in combination with cyclophosphamide (600 mg/m²), administered by intravenous infusion every 21 days (Q3W), for a total of 4 cycles.
  The EC phase commences upon completion of the T phase.
  Immunotherapy Regimen:
  Sintilimab (200 mg), administered by intravenous infusion every three weeks (Q3W).
  Dosing begins on Day 2 of the chemotherapy cycles, for a total of 8 treatment cycles.
  Interventions: Drug: Neoadjuvant Chemotherapy (NACT); Drug: Immunotherapy (Sintilimab)
- Chemotherapy + Immunotherapy + Radiotherapy (Experimental): Neoadjuvant chemotherapy combined with immunotherapy（same as Arm1) + Neoadjuvant Radiotherapy
  Interventions: Radiation: Neoadjuvant radiotherapy; Drug: Neoadjuvant Chemotherapy (NACT); Drug: Immunotherapy (Sintilimab)

INTERVENTIONS:
Radiation: Neoadjuvant radiotherapy — Neoadjuvant Radiotherapy Regimen:
  1. Radiotherapy Technique: Stereotactic Body Radiation Therapy (SBRT) Radiation Dose and Fractionation: 8 Gy per fraction, for a total of 3 fractions, amounting to a total dose of 24 Gy
  2. Radiotherapy Schedule: Irradiation begins on the second day of the first chemotherapy cycle and is administered every other day
  3. Target Volume Definition: The radiotherapy target volume is defined based on baseline imaging (e.g., CT, MRI, or PET-CT)
  4. Radiotherapy Equipment and Planning: Treatment is delivered using a linear accelerator equipped with Image-Guided Radiotherapy (IGRT) technology to ensure precise irradiation and dose optimization
  Arms: Chemotherapy + Immunotherapy + Radiotherapy
Drug: Neoadjuvant Chemotherapy (NACT) — Neoadjuvant Chemotherapy Regimen:
  A sequential chemotherapy strategy is adopted, with the specific regimen as follows:
  Taxane-based Chemotherapy Phase (T Phase):
  Nab-paclitaxel (125 mg/m²), administered by intravenous infusion on Day 1 and Day 8 of each 21-day cycle (Q3W), for a total of 4 cycles.
  Anthracycline-based Combination Chemotherapy Phase (EC Phase):
  Epirubicin (75-100 mg/m²) in combination with cyclophosphamide (600 mg/m²), administered by intravenous infusion every 21 days (Q3W), for a total of 4 cycles.
  The EC phase commences upon completion of the T phase.
Drug: Immunotherapy (Sintilimab) — Immunotherapy Regimen:
  Sintilimab (200 mg), administered by intravenous infusion every three weeks (Q3W).
  Dosing begins on Day 2 of the chemotherapy cycles, for a total of 8 treatment cycles.

SUMMARY:
This study is a prospective, randomized controlled clinical trial designed to evaluate the efficacy and safety of combining radiotherapy, chemotherapy, and immunotherapy in the neoadjuvant treatment of high-risk HR+/HER2- breast cancer patients.

The study plans to enroll treatment-naïve HR+/HER2- breast cancer patients aged 18-75 with high-risk features (e.g., tumor size ≥3 cm or lymph node positivity, Ki-67 ≥20%). Eligible subjects will be randomized in a 1:1 ratio into two groups: the control group will receive neoadjuvant chemotherapy (nab-paclitaxel followed by epirubicin + cyclophosphamide) in combination with sintilimab immunotherapy; the experimental group will receive the same chemotherapy and immunotherapy regimen with the addition of stereotactic body radiotherapy (SBRT) administered early during treatment, at a prescribed dose of 8 Gy per fraction for 3 fractions, with one fraction per day.

The study has dual primary endpoints: pathological complete response (pCR,) and objective response rate (ORR ). Secondary endpoints include 3-year event-free survival (EFS), incidence of adverse events (CTCAE v5.0), and postoperative cosmetic outcomes of the breast. The study design incorporates hierarchical testing to control for multiplicity, and long-term follow-up is planned to evaluate survival benefits.

The study has been approved by the ethics committee, and all participants are required to provide written informed consent. The results are expected to offer a novel neoadjuvant treatment strategy for high-risk HR+/HER2- breast cancer patients and improve their therapeutic outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed, untreated breast cancer;
2. Age: 18 years ≤ age ≤ 75 years;
3. Histologically confirmed hormone receptor-positive (HR+) tumor specimen (estrogen receptor [ER] ≥ 10%);
4. Human epidermal growth factor receptor-2 immunohistochemistry (HER2-IHC) result of 0/1+ or 2+ with negative fluorescence in situ hybridization (FISH) test;
5. Histologically confirmed cell proliferation index (Ki67) ≥ 20%;
6. Programmed death-ligand 1 combined positive score (PD-L1 CPS) evaluable (i.e., availability of fresh/archived specimens);
7. Good pulmonary function;
8. Adequate hepatic and renal function;
9. Histological grade ≥ 2;
10. cN0, cT ≥ 3 cm or cN1-3, cT ≥ 2 cm (cT: clinically assessed maximum diameter of primary tumor; cN: clinically assessed regional lymph node status);
11. Eastern Cooperative Oncology Group Performance Status (ECOG score) 0-1. Exclusion Criteria:

1.Pregnancy; 2.Tumor > 8 cm with skin ulceration; 3.History of thoracic radiotherapy or contraindications to radiotherapy; 4.Active autoimmune disease; 5.Prior use of PD-L1 antibody therapy; 6.De novo breast cancer; 7.There are factors that may significantly increase the risk of lung or cardiac toxicity related to radiotherapy, such as (1) maximum lung depth(MLD) >3.2cm； (2) maximum heart distance(MHD) <2.4cm。

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate（pCR） | Pathological diagnosis results were obtained tithin one month after the operation
  Postoperative pathological assessment (tumor Miller-Payne system grading and axillary lymph node pathological assessment)

SECONDARY OUTCOMES:
Objective response rate(ORR) | At the end of Cycle 8 (each cycle is 28 days)
  The proportion of patients achieving complete response (CR) and partial response (PR) after tumor treatment was used as the second endpoint of the primary endpoint for hierarchical testing.
Event-free survival rate | Long-term follow-up monitoring was conducted until 3 years after enrollment
  The time from randomization to the event (recurrence, metastasis or death)
Incidence of adverse reactions | 1 year
  Continuous monitoring, assessment and patient feedback.

OTHER OUTCOMES:
The breast-conserving rate of breast malignant tumor surgery | Perioperative/Periprocedural
  The breast-conserving rate of breast malignant tumor surgery

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No